CLINICAL TRIAL: NCT05383326
Title: Longitudinal Analysis of the Vaginal Microbiome
Status: Completed | Type: Observational
Sponsor: Viome (Industry)
Responsible Party: Sponsor
Other Study IDs: V174
Record Dates: First submitted 2022-05-16; First posted 2022-05-20 (Actual); Last update posted 2023-12-12 (Actual); Status verified 2023-12

CONDITIONS: Vaginal Microbiome
Keywords: vaginal pH; vaginal microbiome; menstrual cycle

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This is a longitudinal, observational study with the goal of understanding vaginal microbiome changes both within a single day and across a menstrual cycle. The study will be composed of at least 10 women that have regular menstrual cycles and are 18 years of age or older. This study is direct to participant and will NOT utilize clinical sites.

DETAILED DESCRIPTION:
Eligible women will be recruited into the study. They will be consented and asked to complete a health questionnaire. On six separate days during two menstrual cycles, they will be asked to collect vaginal swab samples (total of 12). For each sample collection, they will answer the sample collection questionnaire. Samples will be returned to Viome labs for analysis.

ELIGIBILITY:
Inclusion Criteria:

* Biological sex is female
* Willing to collect own vaginal samples
* Willing to answer health questions
* Experience menstrual cycles regularly (a monthly cycle)

Exclusion Criteria:

* Pregnant
* Antibiotic use in the past 3 months

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: At least 10 women with regular menstrual cycles age 18 or older that meet the inclusion criteria.
Sampling Method: Non-Probability Sample
Enrollment: 29 (Actual)
Dates: Start 2022-07-07 (Actual); Primary Completion 2023-08-20 (Actual); Study Completion 2023-08-20 (Actual)

PRIMARY OUTCOMES:
Identification of vaginal microbial taxonomy | 1 year
  A vaginal metatranscriptomic test will be used to analyze the vaginal microbiome taxonomy
Identification of vaginal microbial functions | 1 year
  A vaginal metatranscriptomic test will be used to analyze the vaginal microbiome functions

CONTACTS AND LOCATIONS:
Overall Officials: Momchilo Vuyisich, Principal Investigator — Viome; Guruduth Banavar, Principal Investigator — Viome
Locations (1):
- Viome Life Sciences, Bothell, Washington, United States